CLINICAL TRIAL: NCT02022904
Title: Development of a Novel Method to Detect Prostate Cancer Circulating Tumor Cells (CTCs) Based on Epithelial-mesenchymal Transition Biology
Brief Title: Prostate Cancer Circulating Tumor Cells Based on Epithelial-Mesenchymal Transition Biology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00037349
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; metastatic; castrate resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metastatic prostate cancer (Experimental): Near infrared (NIR) emissive nanotechnology
  Interventions: Device: Near infrared (NIR) emissive nanotechnology

INTERVENTIONS:
Device: Near infrared (NIR) emissive nanotechnology

SUMMARY:
This is a minimal risk correlative clinical blood-drawing protocol. The objective of this lead in pilot component is to determine whether Circulating Tumor Cells (CTC's) can be captured using the novel mesenchymal-marker based Near Infrared-Emissive Polymersomes (NIR-EPs), the PSMA-based NIR-EP, and the epithelial EpCAM-based NIR-EP. If successful, the capture method will be evaluated further in the larger comparative study.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of adenocarcinoma of the prostate
* Clinical or radiographic evidence of metastatic disease
* Evidence of disease progression on androgen deprivation therapy (ADT) as evidenced by either of the following in the past:

  1. Two consecutive PSA levels greater than the PSA nadir achieved on ADT, separated by greater than one week
  2. Radiographic evidence of disease progression as defined by new bone scan lesions or soft tissue/visceral metastases >2 cm in diameter.
  3. Clinical progression as determined by the treating physician.
* Age greater than 18 years.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of intercurrent or past medical or psychiatric illness that would make participation in a blood drawing protocol difficult or not feasible at the discretion of the principal investigator or co-investigator(s)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Non-detection rate of CTC's in men with CRPC | at baseline, month 3, and progression (up to 18 months)
  Non-detection rate of CTC's in men with CRPC will be measured at baseline, month 3, and at progression

SECONDARY OUTCOMES:
Median number of CTC's detected by each capture method | baseline, month 3, and progression (up to 18 months)
  Calculate for each patient the number of CTC's detected by each capture method (novel and standard).
Change in median number of CTC's for each method | at baseline, month 3, and progression (up to 18 months)
  For each method, we will plot the change across time (baseline, cycle 3, and at progression) in the median number of CTC's for each method (novel and standard).
Correlation of CTC enumeration with presenting clinical stage | at baseline, month 3, and progression (up to 18 months)
Correlation of CTC enumeration with sites of metastatic disease | at baseline, month 3, and progression (up to 18 months)
Correlation of CTC enumeration with Gleason sum | at baseline, month 3, and progression (up to 18 months)
Correlation of CTC enumeration with PSA kinetics | at baseline, month 3, and progression (up to 18 months)
Correlation of CTC enumeration with therapies | at baseline, month 3, and progression (up to 18 months)
Correlation of CTC enumeration with overall survival | at baseline, month 3, and progression (up to 18 months)
Correlation of CTC enumeration with progression-free survival | at baseline, month 3, and progression (up to 18 months)
Correlation of CTC enumeration with response to therapy | at baseline, month 3, and progression (up to 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, Principal Investigator — Duke University